CLINICAL TRIAL: NCT04250350
Title: An Open-Label, Single-Arm Study to Assess the Safety and Efficacy of Lebrikizumab in Adolescent Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Study to Assess the Safety and Efficacy of Lebrikizumab (LY3650150) in Adolescent Participants With Moderate-to-Severe Atopic Dermatitis
Acronym: ADore
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Dermira, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17804; J2T-DM-KGAE (Other: Eli Lilly and Company); DRM06-AD17 (Other: Dermira, Inc); 2019-004301-28 (EudraCT Number)
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Results first posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-01

CONDITIONS: Atopic Dermatitis
Keywords: Eczema; Dermatitis; Dermatitis, Atopic; Skin Diseases
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis; Skin Diseases | interventions — lebrikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lebrikizumab 250 mg (Experimental): Participants received two subcutaneous (SC) injections of 250 milligram(mg) Lebrikizumab at Baseline and Week 2 followed by a single injection every 2 weeks (Q2W) from Week 4 up to (but not including) Week 52.
  Interventions: Biological: Lebrikizumab

INTERVENTIONS:
Biological: Lebrikizumab — Subcutaneous injection
  Other Names: LY3650150; DRM06

SUMMARY:
This is an open-label, single arm study of 52 weeks duration. The study will assess the safety and efficacy of lebrikizumab in adolescent participants (≥12 to <18 years weighing ≥40 kilograms) with moderate-to-severe atopic dermatitis (AD) who are candidates for systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adolescent (≥12 years to <18 years, and weighing ≥40 kg).
2. Chronic AD (according to American Academy of Dermatology Consensus Criteria) that has been present for ≥1 year before the screening visit.
3. Eczema Area and Severity Index (EASI) score ≥16 at the baseline visit.
4. Investigator Global Assessment (IGA) score ≥3 (scale of 0 to 4) at the baseline visit
5. ≥10% body surface area (BSA) of AD involvement at the baseline visit.
6. History of inadequate response to treatment with topical medications; or determination that topical treatments are otherwise medically inadvisable.

Exclusion Criteria:

1. Participation in a prior lebrikizumab clinical study.
2. Treatment with the following prior to the baseline visit:

   1. An investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer.
   2. Dupilumab within 8 weeks.
   3. B-cell-depleting biologics, including to rituximab, within 6 months.
   4. Other biologics within 5 half-lives (if known) or 16 weeks, whichever is longer.
3. Treatment with a live (attenuated) vaccine within 12 weeks of the baseline visit or planned during the study.
4. Uncontrolled chronic disease that might require bursts of oral corticosteroids.
5. Evidence of active acute or chronic hepatitis
6. History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening.
7. History of malignancy, including mycosis fungoides, within 5 years before the screening visit, except completely treated in situ carcinoma of the cervix, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin.
8. Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 206 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (70):
- United States (48):
  - Pinnacle Research Group, Anniston, Alabama
  - Arkansas Research Trials, LLC, North Little Rock, Arkansas
  - Hope Clinical Research, Canoga Park, California
  - First OC Dermatology, Fountain Valley, California
  - MD Studies, Fountain Valley, California
  - Integrative Skin Science and Research, Sacramento, California
  - University of California, San Diego/Rady Children's Hospital, San Diego - Pediatric & Adolescent Dermatology, San Diego, California
  - Southern California Dermatology, Inc., Santa Ana, California
  - IMMUNOe International Research Centers, Centennial, Colorado
  - C&R Research Services USA, Coral Gables, Florida
  - Florida Academic Centers Research and Education, LLC, Coral Gables, Florida
  - Pediatric Skin Research, LLC, Coral Gables, Florida
  - Encore Medical Research, Hollywood, Florida
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - Well Pharma Medical Research Corp., Miami, Florida
  - Sanchez Clinical Research Inc, Miami, Florida
  - Miami Dermatology and Laser Research, Miami, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Georgia Pollens Clinical Research Centers, Inc, Albany, Georgia
  - Advanced Medical Research, Sandy Springs, Georgia
  - Georgia Skin & Cancer Clinic, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - Sneeze, Wheeze, & Itch Associates LLC, Normal, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Kansas Medical Clinic, Topeka, Kansas
  - Skin Sciences, PLLC, Louisville, Kentucky
  - Tulane Univ School of Med, New Orleans, Louisiana
  - Dermatology and Skin Cancer Specialists, Rockville, Maryland
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - St Joseph Dermatology and Vein Clinic, Saint Joseph, Michigan
  - Central Dermatology PC, St Louis, Missouri
  - ALLCUTIS Research, Portsmouth, New Hampshire
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Advanced Asthma and Allergy, Watertown, New York
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Central States Research, Tulsa, Oklahoma
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Paddington Testing Company Inc, Philadelphia, Pennsylvania
  - Arlington Research Center, Inc, Arlington, Texas
  - Encore Imaging & Medical Research, Houston, Texas
  - Cutis Wellness Dermatology, Laredo, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Acclaim Dermatology, PLLC, Sugar Land, Texas
  - Center for Clinical Studies, Webster, Texas
  - PI-Coor Clinical Research, LLC, Burke, Virginia
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Australia (8):
  - Woden Dermatology, Phillip, Australian Capital Territory
  - The Skin Hospital, Sydney, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - Sinclair Dermatology, East Melbourne, Victoria
  - Royal Childrens Hospital Melbourne, Parkville, Victoria
  - Burswood Dermatology, Victoria Park, Western Australia
  - Captain Stirling Medical Centre, Nedlands
- Canada (5):
  - Institute for Skin Advancement, Calgary, Alberta
  - CARe Clinic, Red Deer, Alberta
  - Lynderm Research Inc., Markham, Ontario
  - The Centre for Clinical Trials, Inc, Oakville, Ontario
  - AvantDerm, Toronto, Ontario
- Poland (9):
  - Grazyna Pulka Specjalistyczny Osrodek "ALL-MED", Krakow, Lesser Poland Voivodeship
  - Diamond Clinic, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Evimed, Warsaw, Masovian Voivodeship
  - Zespol Naukowo - Leczniczy "Iwolang" Sp. z o.o., Iwonicz-Zdrój, Podkarpackie Voivodeship
  - Provita Sp. z o.o, Katowice
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 w Lublinie, Lublin
  - CityClinic Przychodnia Lekarsko-Psychologiczna, Wroclaw
  - Dermoklinika Centrum Medyczne s.c. M. Kierstan J. Narbutt A. Lesiak, Lodz, Łódź Voivodeship
  - Gabinet Dermatlogiczny. Beata Krecisz, Kielce, Świętokrzyskie Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Paller AS, Flohr C, Eichenfield LF, Irvine AD, Weisman J, Soung J, Pinto Correia A, Natalie CR, Rodriguez Capriles C, Pierce E, Reifeis S, Gontijo Lima R, Armengol Tubau C, Laquer V, Weidinger S. Safety and Efficacy of Lebrikizumab in Adolescent Patients with Moderate-to-Severe Atopic Dermatitis: A 52-Week, Open-Label, Phase 3 Study. Dermatol Ther (Heidelb). 2023 Jul;13(7):1517-1534. doi: 10.1007/s13555-023-00942-y. Epub 2023 Jun 15. PMID 37318750
- See also: Study to Assess the Safety and Efficacy of Lebrikizumab (LY3650150) in Adolescent Participants With Moderate-to-Severe Atopic Dermatitis (ADore) — https://trials.lillytrialguide.com/en-US/trial/3TxlZTL9UMFNAZAnnCFnbk

RESULTS

PARTICIPANT FLOW:
Groups:
- Lebrikizumab 250 mg: Participants received two subcutaneous (SC) injections of 250 mg Lebrikizumab at Baseline and Week 2 followed by a single injection every 2 weeks (Q2W) from Week 4 up to (but not including) Week 52.
Period: Overall Study
Arm/Group | Lebrikizumab 250 mg
Started | 206
Completed | 172
Not Completed | 34
Not completed — Withdrawal by Subject | 13
Not completed — Lost to Follow-up | 8
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 4
Not completed — Physician Decision | 1
Not completed — Participant moved out of the country/non-compliance | 3

BASELINE CHARACTERISTICS:
Population: All enrolled or randomized participants who received at least one dose of study drug.
Groups:
- Lebrikizumab 250 mg: Participants received 250 mg Lebrikizumab SC at baseline and Week 2. From Week 4 onwards, all participants received 250 mg lebrikizumab SC every 2 weeks up to (but not including) Week 52.
Arm/Group | Lebrikizumab 250 mg
Number analyzed (Participants) | 206
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 206
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (1.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 24
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 26
  White | 138
  More than one race | 11
  Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 20
  United States | 111
  Poland | 63
  Australia | 12
Weight [Count of Participants; unit: Participants]
  <60 kg | 92
  >=60 - <100 kg | 95
  >= 100 kg | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Discontinued From Study Treatment Due to Adverse Events (AEs)
Description: The percentage of participants who discontinued from study treatment due to 1 or more AEs assessed is summarized cumulatively. A summary of all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Week 52
Population: All enrolled participants.
Measure: Number; unit: percentage of participants
Groups:
- Lebrikizumab 250 mg: Participants received two SC injections of 250 mg Lebrikizumab at Baseline and Week 2 followed by a single injection Q2W from Week 4 up to (but not including) Week 52.
Arm/Group | Lebrikizumab 250 mg
Number analyzed (Participants) | 206
percentage of participants | 2.4

2. Secondary Outcome: Percentage of Participants With an Investigator Global Assessment (IGA) Score of 0 or 1 and a Reduction ≥2-points From Baseline
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: Week 52
Population: All participants with evaluable data for IGA score of 0 or 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250 mg
Number analyzed (Participants) | 206
percentage of participants | 62.6 [55.6 to 69.6]

3. Secondary Outcome: Percentage of Participants Achieving ≥75% Reduction From Baseline in Eczema Area and Severity Instrument (EASI) Score (EASI-75)
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  The EASI responder is defined as a participant who achieves a ≥ 75% improvement from baseline in the EASI score.
Time Frame: Week 52
Population: All participants with evaluable data for EASI-75.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250 mg
Number analyzed (Participants) | 206
percentage of participants | 81.9 [76.5 to 87.4]

4. Secondary Outcome: Percentage Change From Baseline in EASI Score
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
Time Frame: Baseline, Week 52
Population: All participants with evaluable data for EASI score.
Measure: Mean (95% Confidence Interval); unit: percentage change
Groups:
- Lebrikizumab 250 mg: Participants received two SC injections of 250 mg Lebrikizumab at Baseline and Week 2 followed by a single injection Q2W from Week 4 through Week 52.
Arm/Group | Lebrikizumab 250 mg
Number analyzed (Participants) | 206
percentage change | -86.0 [-89.1 to -83.0]

5. Secondary Outcome: Percentage of Participants Achieving EASI-50 (≥50 Reduction From Baseline in EASI Score)
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  The EASI responder is defined as a participant who achieves a ≥ 50% improvement from baseline in the EASI score.
Time Frame: Week 52
Population: All participants with evaluable data for EASI-50.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250 mg
Number analyzed (Participants) | 206
percentage of participants | 94.4 [91.1 to 97.7]

6. Secondary Outcome: Percentage of Participants Achieving EASI-90 (≥90% Reduction From Baseline in EASI Score)
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  The EASI responder is defined as a participant who achieves a ≥ 90% improvement from baseline in the EASI score.
Time Frame: Week 52
Population: All participants with evaluable data for EASI-90.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250 mg
Number analyzed (Participants) | 206
percentage of participants | 61.4 [54.5 to 68.3]

7. Secondary Outcome: Change From Baseline in Body Surface Area (BSA)
Description: The BSA affected by AD will be assessed for 4 separate body regions: head and neck, trunk (including genital region), upper extremities, and lower extremities (including the buttocks). Each body region will be assessed for disease extent ranging from 0% to 100% involvement. BSA was calculated using the participant's palm using the 1% rule, 1 palm was equivalent to 1% with estimates of the number of palms it takes to cover the affected AD area. Maximum number of palms were 10 palms for head and neck (10%), 20 palms for upper extremities (20%), 30 palms for trunk, including axilla and groin (30%), 40 palms for lower extremities, including buttocks (40%). Percent of BSA for a body region was calculated as = total number of palms in a body region * % surface area equivalent to 1 palm. Overall percent BSA of all 4 body regions ranges from 0% to 100 % with higher values representing greater severity of AD.
Time Frame: Baseline, Week 52
Population: All participants with evaluable data for BSA.
Measure: Mean (Standard Deviation); unit: percentage of body surface area
Arm/Group | Lebrikizumab 250 mg
Number analyzed (Participants) | 172
percentage of body surface area | -37.63 (21.071)

8. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Information System (PROMIS) Anxiety
Description: PROMIS® is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. Participants ≤17 years will complete pediatric versions for the duration of the study. PROMIS anxiety has 8 questions on Emotion Distress-Anxiety (or Pediatric Anxiety Symptom). Each question has 5 response options with values from 1 to 5. Total raw scores were converted to T-Scores (mean = 50 and a standard deviation = 10) with higher scores representing greater anxiety.
Time Frame: Baseline, Week 52
Population: All participants with evaluable data for PROMIS Anxiety.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Lebrikizumab 250 mg
Number analyzed (Participants) | 170
T-score | -6.34 (9.979)

9. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Information System (PROMIS) Depression
Description: PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. The PROMIS measures will be completed by the participant in the study clinic. PROMIS depression has 8 questions on Emotion Distress-Depression. Questions are measured on a 5-point scale with 1 being "Never" and 5 being "Always". Responses for each section will be summed and converted to T-Scores using the Assessment Center PROMIS Scoring Service, which rescales the raw score to a standardized T-Score with a population mean of 50 and a standard deviation of 10. Total raw scores were converted to T-scores with higher scores indicating greater severity of symptoms.
Time Frame: Baseline, Week 52
Population: All participants evaluable data for PROMIS Depression.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Lebrikizumab 250 mg
Number analyzed (Participants) | 169
T-score | -3.43 (9.057)

10. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI)
Description: The DLQI questionnaire designed for participants aged 17 years or more is a 10-item, validated questionnaire used to assess the impact of skin disease on the quality of life of an affected person. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment, over the previous week. Response categories include "Not at all," "A little," "A lot," and "Very much," with corresponding scores of 0, 1, 2, and 3 respectively. Questions 3-10 also have an additional response category of "Not relevant" which is scored as "0". Questions are scored from 0 to 3, giving a possible total score range from 0 (no impact of skin disease on quality of life) to 30 (maximum impact on quality of life). A high score is indicative of a poor quality of life.
Time Frame: Baseline, Week 52
Population: All participants with evaluable data for DLQI.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lebrikizumab 250 mg
Number analyzed (Participants) | 35
score on a scale | -8.92 [-10.8 to -7.1]

11. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI)
Description: The CDLQI questionnaire is designed for use in children (4 to 16 years of age). It consists of 10 items that are grouped into 6 domains: symptoms & feelings, leisure, school or holidays, personal relationships, sleep, & treatment. The scoring of each question is: Very much =3; Quite a lot = 2; Only a little = 1; Not at all = 0. CDLQI total score is calculated by summing all 10 items responses and has a range of 0 to 30 (higher scores are indicative of greater impairment).
Time Frame: Baseline, Week 52
Population: All participants with evaluable data for CDLQI.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Lebrikizumab 250 mg
Number analyzed (Participants) | 168
score on a scale | -6.45 [-7.4 to -5.5]

12. Secondary Outcome: Pharmacokinetics (PK): Average Serum Concentration of Lebrikizumab
Description: Pharmacokinetics (PK): Average Serum Concentration of Lebrikizumab was evaluated at Week 52.
Time Frame: Predose: Week 52
Population: All participants with evaluable PK data at Week 52.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (μg/mL)
Arm/Group | Lebrikizumab 250 mg
Number analyzed (Participants) | 138
microgram per milliliter (μg/mL) | 82.3 (39.8)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- Lebrikizumab 250mg: Participants received two SC injections of 250 mg Lebrikizumab at Baseline and Week 2 followed by a single injection Q2W from Week 4 up to (but not including) Week 52.
Arm/Group | Lebrikizumab 250mg
All-Cause Mortality (participants affected / at risk) | 1/206
Serious Adverse Events (participants affected / at risk) | 5/206
Other Adverse Events (participants affected / at risk) | 133/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Lebrikizumab 250mg (N=206)
Cardiac arrest (Cardiac disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1)
Testicular torsion (Reproductive system and breast disorders) | 1/98 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Lebrikizumab 250mg (N=206)
Eosinophilia (Blood and lymphatic system disorders) | 8 (9)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Sinus arrhythmia (Cardiac disorders) | 1 (1)
Thyroglossal cyst (Congenital, familial and genetic disorders) | 1 (1)
Type v hyperlipidaemia (Congenital, familial and genetic disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Atopic keratoconjunctivitis (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (3)
Conjunctivitis allergic (Eye disorders) | 4 (8)
Episcleritis (Eye disorders) | 1 (1)
Eye irritation (Eye disorders) | 1 (1)
Eyelids pruritus (Eye disorders) | 2 (2)
Ocular hyperaemia (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Angular cheilitis (Gastrointestinal disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (9)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Toothache (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 3 (5)
Injection site erythema (General disorders) | 2 (3)
Injection site pain (General disorders) | 3 (8)
Injection site reaction (General disorders) | 2 (3)
Malaise (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (4)
Vaccination site erythema (General disorders) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Food allergy (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2)
Multiple allergies (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 10 (12)
Conjunctivitis bacterial (Infections and infestations) | 1 (1)
Covid-19 (Infections and infestations) | 19 (19)
Cystitis (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Eczema herpeticum (Infections and infestations) | 1 (1)
Epididymitis (Infections and infestations) | 1/98 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Herpes dermatitis (Infections and infestations) | 5 (11)
Herpes ophthalmic (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 3 (7)
Hordeolum (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 20 (28)
Oral herpes (Infections and infestations) | 11 (22)
Otitis media (Infections and infestations) | 2 (2)
Paronychia (Infections and infestations) | 3 (5)
Pelvic inflammatory disease (Infections and infestations) | 1/108 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4)
Staphylococcal skin infection (Infections and infestations) | 1 (2)
Tinea versicolour (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 13 (15)
Urinary tract infection (Infections and infestations) | 3 (3)
Wound infection (Infections and infestations) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Nail injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (2)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Mean cell haemoglobin concentration decreased (Investigations) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1)
Platelet count increased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Gluten sensitivity (Metabolism and nutrition disorders) | 1 (1)
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cutaneous t-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 12 (15)
Loss of consciousness (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (3)
Persistent depressive disorder (Psychiatric disorders) | 1 (1)
Social anxiety disorder (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/108 (3)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 2/108 (2)
Menstruation irregular (Reproductive system and breast disorders) | 2/108 (2)
Polymenorrhoea (Reproductive system and breast disorders) | 1/108 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Dandruff (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 26 (38)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 (2)
Milia (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 6 (8)
Hypertension (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT04250350/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT04250350/SAP_001.pdf